CLINICAL TRIAL: NCT03059849
Title: Brief Escalation of Adalimumab Treatment for Prevention of Clinical Relapse in IBD
Acronym: BEAT-IBD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2831
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2017-02

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Temporary increase in adalimumab (Active Comparator)
  Interventions: Drug: Adalimumab
- Continued monitoring as per standard of care (No Intervention)

INTERVENTIONS:
Drug: Adalimumab — Dose of adalimumab will be increased by 40mg every 2 weeks.
  Arms: Temporary increase in adalimumab

SUMMARY:
To examine whether a temporary three month increase in adalimumab dosing will prevent relapse in patients with inflammatory bowel disease in clinical remission who have elevated calprotectin.

DETAILED DESCRIPTION:
Patients using adalimumab for Crohn's disease or ulcerative colitis who are in clinical remission will be followed with fecal calprotectin monitoring every 3 months. Patients with a sustained rise in calprotectin who maintain clinical remission will be offered an opportunity to have an increase in adalimumab for three months. Patients who use the three months of increased adalimumab dosing will be compared to patients who do not use increased dosing to determine if relapse rates differ between these two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 and older with Crohn's disease and ulcerative colitis
2. Patients are in clinical remission according to the last 'Abbvie Care' clinical symptom assessment (using Partial Mayo score < 2 or Harvey-Bradshaw Index < 4)
3. Patient using adalimumab at a dose of at least 40mg subcutaneously bi-weekly, and at a maximum dose of 40mg subcutaneously weekly (or 80mg subcutaneously bi-weekly).

Exclusion Criteria:

1. Pregnant women or plans for pregnancy within 3 months of study inclusion
2. Abdominal abscess
3. Inability or unwillingness to provide informed consent
4. Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinical relapse | One year
  Clinical relapse will be based on increased clinical symptoms or endoscopic changes requiring use of corticosteroids, addition of an immunomodulator, change to another biologic therapy, or surgery.

IPD SHARING:
Plan to Share IPD: No